CLINICAL TRIAL: NCT05334316
Title: Individualizing Corticosteroid Use in Pneumonia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yewande Odeyemi, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-009032
Record Dates: First submitted 2022-04-04; First posted 2022-04-19 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Group (No Intervention): Usual care as determined by the patient's primary team. Initiation and daily dosing of corticosteroid treatment will be based on clinicians' preference and clinicians.
- Individualized dosing strategy (Experimental): Biomarker guided corticosteroid use. Initiation of corticosteroid will be recommended based on the an individual treatment rule (ITR) and subsequent dosing of corticosteroid will be recommended based on daily CRP values till CRP <50 mg/L.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Administered intravenously or orally based on daily CRP values and CRP corticosteroid dosing algorithm
  Arms: Individualized dosing strategy

SUMMARY:
In this study, researchers propose a unique (individualized) approach to steroid treatment seeking to give the right dose of steroid to the right patient and at the right time. This study seeks to compare usual care to an individualized steroid dosing strategy by testing a marker of inflammation in the blood called C- reactive protein (CRP). The overall goal is to reduce an individual's exposure to steroids and the risk of potential side effects thereby increasing the potential benefit of using steroids to control inflammation in pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult (≥ 18 years) patients.
* Community acquired pneumonia.

Exclusion Criteria:

* Contraindications or unwillingness to use corticosteroids by patient or provider.
* History of adrenal insufficiency, septic shock, or another absolute indication for steroid use.
* Suspected pulmonary vasculitis or other autoimmune pulmonary disorder.
* Positive pregnancy test
* Comfort care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to individual treatment rule and CRP-guided corticosteroid treatment | First 5 days of hospitalization or until hospital discharge (whichever is sooner)
  Number of eligible subjects that adhered to the timely initiation and daily corticosteroid treatment

SECONDARY OUTCOMES:
In-hospital Disease Progression | First 5 days of hospitalization or until hospital discharge (whichever is sooner)
  Progression on the WHO clinical progression scale from 4 to 10
Need for Advanced Respiratory Support | First 5 days of hospitalization or until hospital discharge (whichever is sooner)
  Number of participants to require use of advanced respiratory support (high flow nasal cannula, non-invasive positive pressure ventilation and invasive ventilation)
Advanced respiratory support free days | First 5 days of hospitalization or until hospital discharge (whichever is sooner)
  Number of days without need for high flow nasal cannula, non-invasive positive pressure ventilation and invasive ventilation within 28 days of need for support. Assign 0 if death occurs with 28 days.
ICU and hospital free days | First 5 days of hospitalization or until hospital discharge (whichever is sooner)
  Number of days patient was alive outside the ICU or hospital within the first 28 days of admission
Mortality | First 5 days of hospitalization or until hospital discharge (whichever is sooner)
  Number of subject deaths

CONTACTS AND LOCATIONS:
Overall Officials: Yewande Odeyemi, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20544831